CLINICAL TRIAL: NCT06455436
Title: Dimensional Changes of Peri-implant Tissue in Immediate Implants With Individualized Healing Abutments Using a CAD/CAM Technique: Randomized Controlled Clinical Trial
Brief Title: Dimensional Changes of Peri-implant Tissue in Immediate Implants With Individualized Healing Abutments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2023-10
Record Dates: First submitted 2024-05-30; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Dental Implant; Immediate Dental Implant; Wound Heal
Keywords: implant; soft tissue

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Will receive standard healing abutments
  Interventions: Device: Standard healing abutment
- Individualized healing abutment group (Experimental): Will receive individualized healing abutments
  Interventions: Device: Individualized healing abutment

INTERVENTIONS:
Device: Standard healing abutment — Participants will undergo a surgery to place an immediate klockner dental implant and will be receive a standard healing abutment
  Arms: Control group
Device: Individualized healing abutment — Participants will undergo a surgery to place an immediate klockner dental implant and will be receive an individualized healing abutment
  Arms: Individualized healing abutment group

SUMMARY:
The loss of a tooth leads to a series of biological changes in the tissues, resulting in bone resorption and gingival collapse. To avoid these problems, it has been proposed to place immediate post-extraction implants, allowing a reduction in treatment time and the number of surgeries, as well as better maintenance of the tissues. This technique can be performed with standard abutments after implant placement or, more recently, the use of temporary abutments has been proposed.

DETAILED DESCRIPTION:
Objective: To check if custom healing abutments manufactured using CAD/CAM technique in immediate implants promote greater dimensional stability of the peri-implant tissue compared to standard healing abutments.

Methods: After the extraction, an immediate Klockner Vega+ implant will be placed and the gap will be filled with a bone substitute (Cerabone, Botiss). The patient will then be randomized to the control group (standard healing abutment) or the test group (custom healing abutment using CAD/CAM technique). In the latter case, a peripheral seal is achieved, allowing for wound closure and stabilization of the clot with the same shape as the crown in its transmucosal part.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ( 25 years old).
* Need for extraction of an irrational tooth to be treated in the molar/premolar position of the upper/lower arch.
* Presence of 2mm of keratinized gingiva.
* Bone dehiscence in the alveolar walls of 2 mm. 2 mm.
* Adequate amount of bone in the interradicular septum to stabilize the implant (minimum height 10 mm, minimum width 4 mm at the base of the septum).
* Plaque index (FMSPI, full mouth score plaque index) < 10%.
* Non-smokers or smokers of less than 10 cigarettes per day.
* Absence of systemic diseases that contraindicate implant surgery.

Exclusion Criteria:

* Presence of alveoli with dehiscence >2mm.
* Presence of adjacent implants.
* < 2mm of keratinized gingiva.
* Presence of active infection (fistula, suppuration) at the extraction site.
* Presence of apical granuloma >2mm in diameter in the root(s) of the tooth or teeth to be extracted.
* Residual bone apical to the extraction insufficient to anchor the implant.
* Pregnant or lactating women.
* Severe cognitive or psychiatric disorders.
* Compromised general health status ( ASA IV).
* Use of drugs that alter bone metabolism and healing.
* Absence of manual primary stability of the implant
* Bone dehiscence or fenestration after implant placement (manual rotation).
* Gap 2mm between the implant and the vestibular bone wall.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Buccal-lingual/palatal soft tissue dimensional changes | 12 months
  They will be evaluated after superimposing the initial STL files with the follow-up ones. In addition, photos, periapical radiographs and a new intraoral scan at 3 months, 6 months and 1 year will be taken. In a 2D buccal-lingual slice corresponding to the center of the ridge, measure at the vestibular and palatal level from the point of maximum preoperative STL soft tissue contour (mucosal margin and at 3 mm and 5 mm apical to the margin).

SECONDARY OUTCOMES:
Dehiscence of peri-implant vestibular and lingual/palatal mucosa: | 12 months
  Dehiscence can be assessed by carefully examining the peri- implant mucosa for any signs of tissue separation or exposure. This can be done visually during clinical examination.
Vestibulo-lingual/palatal dimensional changes of the alveolar bone (CBCT) | 12 months
  To measure dimensional changes in the alveolar bone, you can use cone-beam computed tomography (CBCT) scans. Compare CBCT images taken at different time points to quantify any changes in bone dimensions. measure dimensional changes in the alveolar bone, you can use cone-beam computed tomography (CBCT) scans. Compare CBCT images taken at different time points to quantify any changes in bone dimensions.
Horizontal remodeling of vestibular and lingual/palatal cortex (CBCT) | 12 months
  CBCT scans can also be used to assess horizontal remodeling of the cortical bone. Analyze the CBCT images to measure changes in cortical thickness or contour.
Thickness of vestibular and lingual/palatal cortex (CBCT) | 12 months
  CBCT scans can provide measurements of cortical thickness in the vestibular and lingual/palatal regions of the alveolar bone.
Vertical changes of the vestibular and lingual/palatine cortex (CBCT) | 12 months
  Use CBCT scans to measure any vertical changes in the vestibular and lingual/palatal cortical bone regions.
Marginal bone level (periapical x-ray) | 12 months
  Periapical X-rays are commonly used to assess marginal bone levels around dental implants. Measure the distance from the implant-abutment interface to the crestal bone on these radiographs.
Probing pocket depth | 12 months
  Probing pocket depth can be measured using periodontal probes. Insert the probe gently into the peri-implant sulcus and measure the distance from the mucosal margin to the implant-abutment interface.
Bleeding/Suppuration on probing | 12 months
  Assess bleeding or suppuration during probing. Note if there is any bleeding or exudate from the peri-implant sulcus when probing the tissues.
Implant survival | 12 months
  Implant survival can be determined by assessing whether the implant remains in place and functional over the study period. Any implant removals or failures should be documented.
Patient-reported variables (satisfaction, pain) | 12 months
  Subjective assessment of pain intensity and patient satisfaction using a 10-cm visual analog scale. The extremes of the scale are the extreme expressions of pain and discomfort (i.e., no pain and the worst imaginable pain)
  * Type of variable (units): scale (mm).
  * Time of registration: Appointment 4 (surgery), Appointment 5 (follow-up), Appointment 10 (End of study)

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Albertini, PhD, Principal Investigator — Universidad Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No